CLINICAL TRIAL: NCT07401550
Title: Assessment and Prediction of Cardiovascular Health and Disease Risk Using Longitudinal Wearable Biometrics: a Prospective Cohort Study.
Brief Title: Assessment and Prediction of Cardiovascular Health and Disease Risk Using Wearable Biometrics.
Acronym: BEACON-HEART
Status: Recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Beacon Hospital, Ireland (Unknown)
Responsible Party: Principal Investigator, Rory Lambe, Doctoral Researcher, University College Dublin
Other Study IDs: BEA0247
Record Dates: First submitted 2025-12-07; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases (CVD); Cardiovascular Disease Prevention; Cardiovascular Disease Risk Factor; Coronary Artery Disease (CAD)
Keywords: wearables; wearable devices; cardiovascular health; cardiovascular disease; wearable technology; fitbit; fitabase; remote monitoring; cardiovascular disease prevention; cardiovascular risk reduction; digital biomarker; coronary artery disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cardiovascular disease and healthy individuals: A single prospective cohort will be recruited, comprising predominantly individuals with atherosclerotic cardiovascular disease. Patients with mild, moderate and severe ASCVD will be recruited, including patients from cardiac rehabilitation physiotherapy classes and post-operative percutaneous coronary intervention (PCI) patients. A sub-group with good cardiovascular health - without diagnosed cardiovascular disease - will also be recruited as part of this cohort to facilitate analysis across the full spectrum of cardiovascular health and development of statistical models for cardiovascular health assessment.

SUMMARY:
This prospective, observational cohort study will evaluate the associations between wearable-derived biometrics and cardiovascular health, quantified by the American Heart Association's Life's Essential 8 framework, as well as related cardiovascular risk factors. The study aims to determine whether wearable biometrics can support the assessment of cardiovascular health and cardiovascular disease risk, both when used in isolation and in combination with point-of-care assessments.

DETAILED DESCRIPTION:
Participants will be provided with a Fitbit Charge 6 to wear continuously for six-months. These wearable data will be collected via Fitabase (Small Steps Labs LLC) for the duration of the study.

At baseline, mid-point (three months), and end-point (six months), participants will undergo a clinical cardiovascular health assessment and Life's Essential 8 score will be calculated. Life's Essential 8, established by the American Heart Association, is a composite metric comprising four Health Behaviours and four Health Factors, and provides individuals with a score ranging from 0 (poor health) to 100 (optimal health). Life's Essential 8 health tiers are defined as 'Low' (<50), 'Moderate' (50-79), and 'High' (80-100). Alongside Life's Essential 8, during each clinical assessment, four patient-reported outcome measures will be collected: EQ-5D-5L, International Physical Activity Questionnaire, Patient Health Questionnaire 9, and Generalized Anxiety Disorder 7.

Participants will also complete patient-reported outcome measures online once per week for the duration of the study. These include the Modified Wisconsin Upper Respiratory Symptom Scale (WURSS), Alcohol Intake Questionnaire, Single-Item Sleep Quality Scale (SQS), Patient Health Questionnaire 4 (PHQ-4), and the two-item Modified Hooper Questionnaire for stress and fatigue. Once per month they will complete the Pittsburgh Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years, or older
* Internet access
* Possession of a smartphone compatible with the Fitbit mobile app

Exclusion Criteria:

* Pregnancy
* Unstable medical condition
* Inability to provide informed consent
* Mental or cognitive impairment precluding adherence to study protocol
* Smartwatch cannot be worn, (e.g., allergic reactions), or cannot be worn in accordance with manufacturer guidelines (e.g., amputation, dark tattoos at wrist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will primarily include patients with moderate or poor cardiovascular health who have been diagnosed with atherosclerosis and other cardiovascular disease. A smaller proportion of individuals with good cardiovascular health, without diagnosed cardiovascular disease, will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cross-Sectional Association of Wearable Biometrics with Cardiovascular Health | Baseline, Month 3, and Month 6
  The strength and direction of the associations between wearable-derived biometric data (e.g., heart rate, sleep, step count) and cardiovascular health, quantified using Life's Essential 8 score and each of its individual components. Life's Essential 8 is measured on a scale from 0 to 100, with higher scores representing better cardiovascular health. Clinical cardiovascular assessments will be paired with wearable biometric data from a window of ±2 weeks surrounding the clinical visit date.
Longitudinal Association of Changes in Wearable Biometrics with Changes in Cardiovascular Health | Between assessments of cardiovascular health from baseline to Month 3, Month 3 to Month 6, and baseline to Month 6.
  The strength and direction of the association between changes in wearable-derived biometrics and corresponding changes in cardiovascular health, quantified using Life's Essential 8 score and each of its components, assessed over time both within and between individuals. Life's Essential 8 is measured on a scale from 0 to 100, with higher scores representing better cardiovascular health.

SECONDARY OUTCOMES:
Classification Performance for Life's Essential 8 Tier | Baseline, Month 3, Month 6.
  Model classification performance for discriminating between Life's Essential 8 cardiovascular health tiers using wearable-derived biometrics, with and without partial imputation of Life's Essential 8 components which are measurable by point-of-care testing (diet, nicotine use, HbA1c, lipid profile, BMI, blood pressure). Life's Essential 8 tiers are defined as 'Low' (>50), 'Moderate' (50-79), and 'High' (80-100).
Prediction Accuracy of Change in Life's Essential 8 Score | From baseline to Month 3, Month 3 to Month 6, and baseline to Month 6.
  Statistical model performance in estimating the direction and the magnitude of change in Life's Essential 8 score between assessment timepoints, compared with observed scores. A 10-point change in Life's Essential 8 score is clinically significant.
Cross-Sectional Correlation of Wearable Biometrics with Patient-Reported Psychosocial and Behavioural Risk Factors of Cardiovascular Disease | Baseline, Month 3, Month 6.
  The strength and direction of inter-individual correlation between wearable-derived biometric data and patient-reported outcome measures of alcohol intake, sleep, stress and fatigue, illness, anxiety and depression, physical activity, and quality of life.
Longitudinal Correlation of Weekly and Monthly Changes in Wearable Biometrics with Patient-Reported Psychosocial and Behavioural Risk Factors of Cardiovascular Disease | Baseline through Month 6
  The strength and direction of intra-individual correlation between wearable-derived biometric data and patient-reported outcome measures of alcohol intake, sleep, stress and fatigue, illness, anxiety and depression, physical activity, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rory Lambe, Principal Investigator — University College Dublin
Locations (1):
- Beacon Hospital, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No